CLINICAL TRIAL: NCT06583863
Title: Parasitic Infection Flares up the Activity of Ulcerative Colitis; However, Combined Immunomodulatory Therapy With Anti-parasitic Treatment Could Proceed Toward Remission
Brief Title: Parasitic Infections and Ulcerative Colitis: Combining Anti-parasitic and Immunomodulatory Treatments May Achieve Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Heba M. Aboelela, Lecturer of Medical Parasitology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 16-7-2024
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Echinacea extract; Metronidazole; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator)
  Interventions: Drug: Echinacea Extract
- Group I (Active Comparator)
  Interventions: Drug: MetroNIDAZOLE 500 MG Oral Tablet [Flagyl]
- Group II (Active Comparator)
  Interventions: Drug: Echinacea Extract; Drug: MetroNIDAZOLE 500 MG Oral Tablet [Flagyl]

INTERVENTIONS:
Drug: Echinacea Extract — 175 mg of Echinacea extract was provided as an immunlant therapy twice daily.
  Arms: Control Group; Group II
Drug: MetroNIDAZOLE 500 MG Oral Tablet [Flagyl] — 500 mg of metronidazole was provided as an oral tablets twice daily
  Arms: Group I; Group II

SUMMARY:
The study aimed to explore the link between parasitic infections and the severity of ulcerative colitis (UC). 120 UC patients were divided into three groups: those without infection, those with Giardia lamblia infection treated with metronidazole, and those with Giardia infection treated with a combination of metronidazole and E. purpurea. The results revealed that patients with Giardia infections exhibited more severe UC symptoms. All groups experienced improved symptoms following treatment, but the combination therapy group demonstrated the most significant improvement. Remission rates were highest in the group without infection and the group receiving combination therapy. Additionally, the study identified E. purpurea therapy and a substantial reduction in SCCAI score as significant predictors of higher remission rates.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative Colitis patients had active disease,
* Patients had parasitic infection by G. lambellia,
* Patients free of parasitic infection,
* Patients free of exclusion criteria..

Exclusion Criteria:

* Patients had Inflammatory Bowel Disease other than Ulcerative Colitis,
* Patients had multiple parasitic infections,
* Patients had infection by parasites other than G. lambellia,
* Patients who were maintained on immunosuppressant therapy,
* Patients who were in remission and patients refused to sign the written consent to participate in the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% increase in the remission rate of parasitic infection (measured by changes in Serum CRP, Fecal calprotectin, and on the Simple Clinical Colitis Activity Index[SCCAI]) in patients with Ulcerative colitis. | 4 weeks
  Patients had parasitic infection showed significantly higher pre-treatment SCCAI score and FCP level than patients free of infection. Post-treatment SCCAI scores of all patients were significantly lower than the pre-treatment scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha faculty of Medicine, Banhā, El Qalyoubia, Egypt